CLINICAL TRIAL: NCT04162587
Title: Association Between Extracranial Carotid & Intracranial Arterial Stenosis in Ischemic Stroke Patients: Predictors & Outcome
Brief Title: Extracranial Carotid & Intracranial Arterial Stenosis in Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 4
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Ischemic Stroke; Carotid Stenosis
Keywords: Ischemic Stroke; carotid stenosis
MeSH Terms: conditions — Ischemic Stroke; Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1)Patients with significant carotid stenosis only: Patients with significant carotid stenosis without intracranial stenosis.
  Interventions: Other: Carotid duplex+/- MRA neck; Other: brain MRA+/-CT angio on carotid and brain; Other: MRI brain; Other: DSA (digital subtraction angiography)
- 2) Patients with carotid and intracranial stenosis.: Patients with carotid and intracranial stenosis.
  Interventions: Other: Carotid duplex+/- MRA neck; Other: brain MRA+/-CT angio on carotid and brain; Other: MRI brain; Other: DSA (digital subtraction angiography)
- 3) Patients with lone intracranial stenosis.: Patients with lone intracranial stenosis.
  Interventions: Other: Carotid duplex+/- MRA neck; Other: brain MRA+/-CT angio on carotid and brain; Other: MRI brain; Other: DSA (digital subtraction angiography)
- 4) Patients with no significant stenosis: Patients with no significant carotid or intracranial stenosis.
  Interventions: Other: Carotid duplex+/- MRA neck; Other: brain MRA+/-CT angio on carotid and brain; Other: MRI brain

INTERVENTIONS:
Other: Carotid duplex+/- MRA neck — Carotid duplex and or MRA neck
Other: brain MRA+/-CT angio on carotid and brain — brain MRA and or CT angiography on carotid and brain
Other: MRI brain — MRI brain with diffusion to detect asymptomatic stroke
Other: DSA (digital subtraction angiography) — DSA (digital subtraction angiography) in some cases to confirm diagnosis.
  Groups: 1)Patients with significant carotid stenosis only; 2) Patients with carotid and intracranial stenosis.; 3) Patients with lone intracranial stenosis.

SUMMARY:
The aim of the work is to; elucidate how the presence of carotid stenosis influence the pattern of stroke and also how it interact with other risk factors for stroke. Also identify predictors of intracranial stenosis and outcome in patients with carotid stenosis with or without intracranial stenosis.

DETAILED DESCRIPTION:
Patients:

Ischemic stroke patients admitted to Neurology department in Mansoura University hospital (MUH) will be studied

The patients will be grouped as follow:

1. Patients with significant carotid stenosis without intracranial stenosis.
2. Patients with carotid and intracranial stenosis.
3. Patients with lone intracranial stenosis.
4. patients with no significant carotid or intracranial stenosis.

Methods:

Studied patients will undergo the following:

* Clinical assessment with NIH scale with is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit, Modified Rankin Scale, Arabic version of Montereal Coginitive Assessment and Arabic version of Beck's Depression Inventory at presentation and after 6 months.
* carotid duplex+/- MRA neck and brain MRA+/-CT angio on carotid and brain (at 0day) and 6m after.
* MRI brain with diffusion to detect asymptomatic stroke at 0 day and 6 months later.
* DSA (digital subtraction angiography) in some cases to confirm diagnosis.
* Laboratory investigations: complete blood count, liver function and renal function tests, random blood sugar, lipid profile.

All patients will be treated with acetyle-salicylic acid(150/day) +/-clopidogrel (75mg /day) +/- statins, plus modification of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Carotid TIA (transient ischemic attack) it should, however, be focal and usually motor-sensory to implicate the carotid artery system or ischemic stroke involving carotid territory.
* Asymptomatic patients with carotid stenosis or anterior circulation stenosis discovered accidentally during investigations for further risk factors.

Exclusion Criteria:

* Major functional impairment (Modified Rankin Scale >/= 3)
* Significant cognitive impairment.
* Contraindication to acetylsalicylic or dual antiplatelet.
* Renal dysfunction precluding safe contrast medium administration.
* pregnancy or refusal.
* Intracranial aneurysm or AVM.
* Intra cerebral hemorrhage or hemorrhagic infarction.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 141 patients of acute ischemic stroke presented by carotid TIA (transient ischemic attack) or asymptomatic patients with carotid stenosis or anterior circulation stenosis discovered accidentally during investigations for further risk factors.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | 24 hours
  The National Institutes of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. The higher score indicate poor outcome.

SECONDARY OUTCOMES:
The modified Rankin Scale | 24 hours
  The modified Rankin Scale is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials. The higher score indicate poor outcome.
Beck's Depression Inventory | 24hours
  The Beck Depression Inventory, created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke. 1988 Dec;19(12):1497-500. doi: 10.1161/01.str.19.12.1497. PMID 3201508
- [Result] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Result] Josephson SA, Hills NK, Johnston SC. NIH Stroke Scale reliability in ratings from a large sample of clinicians. Cerebrovasc Dis. 2006;22(5-6):389-95. doi: 10.1159/000094857. Epub 2006 Aug 4. PMID 16888381
- [Result] Lee SJ, Cho SJ, Moon HS, Shon YM, Lee KH, Kim DI, Lee BB, Byun HS, Han SH, Chung CS. Combined extracranial and intracranial atherosclerosis in Korean patients. Arch Neurol. 2003 Nov;60(11):1561-4. doi: 10.1001/archneur.60.11.1561. PMID 14623728
- [Result] Loftus CM, Harbaugh RE, Fleck JD, Biller J. Carotid occlusive disease: natural history and medical management. In: Winn HR, ed. Youman's Neurological Surgery. 6th ed. Philadelphia, PA: WB Saunders; 2011:3616.
- [Result] Pinzon R, Asanti L, Sugianto, Widyo K. Risk factors of intracranial stenosis among older adults with acute ischemic stroke. unversa Medicinia 2009;28:1-7.
- [Result] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Result] Sayed A, Ahmed S M, Abdelalim A M, Nagah M, Khairy H. Is peripheral arterial disease associated with carotid artery disease in Egyptians? A pilot study. The Egyptian Journal of Neurology, Psychiatry and neurosurgery 2016;53:12-18.
- [Result] Sung YF, Lee JT, Tsai CL, Lin CC, Hsu YD, Lin JC, Chu CM, Peng GS. Risk Factor Stratification for Intracranial Stenosis in Taiwanese Patients With Cervicocerebral Stenosis. J Am Heart Assoc. 2015 Dec 15;4(12):e002692. doi: 10.1161/JAHA.115.002692. PMID 26672078
- [Result] Wong KS, Li H. Long-term mortality and recurrent stroke risk among Chinese stroke patients with predominant intracranial atherosclerosis. Stroke. 2003 Oct;34(10):2361-6. doi: 10.1161/01.STR.0000089017.90037.7A. Epub 2003 Aug 28. PMID 12947158